CLINICAL TRIAL: NCT01740817
Title: A Randomized, Crossover Study to Evaluate the Effect of Lipid Infusion on TLR4 Signaling and Insulin Resistance in Human Muscle
Brief Title: A Study to Evaluate the Effect of Lipid Infusion on Toll Like Receptor 4 (TLR4) Signaling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nicolas Musi, MD, Professor Diabetes Division, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20080015H; 5R01DK080157 (NIH)
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes; Obesity
Keywords: diabetes; obesity; inflammation
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Inflammation | interventions — safflower oil, soybean oil, lecithin emulsion; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intralipid 20%, then saline (Experimental): Participants first received lipid infusion of 30ml/h x48h. After a washout period of 4-6 weeks, they then received saline infusion of 30ml/h x48h.
  Interventions: Drug: Intralipid 20%; Drug: Saline
- Saline, then Intralipid (Experimental): Participants first received saline infusion of 30ml/h x48h. After a washout period of 4-6 weeks, they then received lipid infusion of 30ml/h x48h.
  Interventions: Drug: Intralipid 20%; Drug: Saline

INTERVENTIONS:
Drug: Intralipid 20% — 30 ml/h for 48 h
  Other Names: Liposyn
Drug: Saline — 30 ml/h for 48 h
  Other Names: sodium chloride injection

SUMMARY:
The purpose of this study is to determine whether a lipid infusion can up-regulate toll-like receptor 4 (TLR4) signaling in human subjects

DETAILED DESCRIPTION:
The investigators plan to examine the effect of a lipid infusion on TLR4 expression and insulin sensitivity. A group of 30 subjects aged 18-60 years old, lean (BMI < 26 kg/m2) normal glucose tolerant subjects without a family history of type 2 diabetes will receive a lipid or saline infusion. The subjects will be randomly assigned to first receive either a 48 hour long lipid or saline infusion. Approximately 4-6 weeks later subjects will return to undergo another study (if, in the first study they received lipid, on the second study they will receive saline, and vice versa). A near-equal number of women and men will be included in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have the following laboratory values: Hematocrit ≥ 35%, serum creatinine ≤ 1.5 mg/dl, aspartate aminotransferase (AST) < 2 X upper limit of normal, Alanine aminotransferase (ALT) < 2 X upper limit of normal, alkaline phosphatase < 2 X upper limit of normal, normal urinalysis [no glucose, trace protein, trace ketones, lipase < 50 IU/L, no bacteria, up to 1-3 white blood cells (WBC) and red blood cells (RBC) per hpf], and normal platelets, prothrombin time (PT) and partial thromboplastin time (PTT).
2. Female subjects must be non-lactating. Female patients are eligible only if they have a negative pregnancy test throughout the study period (or postmenopausal). Postmenopausal women taking hormone replacement will be included if they have been on a stable dose for ≥6 months.
3. Subjects whose body weight has been stable (within 2%) for at least three months.

Exclusion Criteria:

1. Subjects with impaired glucose tolerance based on American Diabetes Association criteria.
2. Subjects taking drugs known to affect glucose and lipid homeostasis will be excluded. Statins will be permitted if the subject has been on a stable dose for at least three months. Subjects who have taken for more than a week non-steroidal anti inflammatory drugs (NSAIDS) within two months or systemic steroids, anabolic steroids, growth hormone or immunosuppressants within 12 months will be excluded. Subjects taking low-dose (81 mg/day or less) aspirin will be allowed.
3. Patients with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
4. Recent systemic or pulmonary embolus, impaired renal function, poorly controlled blood pressure (systolic BP>170, diastolic BP>95), resting heart rate >100, electrolyte abnormalities, neuromuscular or musculoskeletal disease.
5. Subjects who smoke.
6. Subjects who engage in a regular exercise program (zero or one exercise sessions per week are allowed).
7. Any subject who has donated blood in the previous two months.
8. Any subject with a hematocrit of less than 35.
9. Subjects who are claustrophobic.
10. Women taking oral contraceptives.
11. alcohol consumption greater than 30 grams daily.
12. baseline plasma triglyceride levels over 200 mg/dl

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD, Principal Investigator — Univerisity of Texas Health Science Center at San Antonio
Locations (1):
- Audie L. Murphy VA Hospital, San Antonio, Texas, United States

REFERENCES:
- [Derived] Hussey SE, Lum H, Alvarez A, Cipriani Y, Garduno-Garcia J, Anaya L, Dube J, Musi N. A sustained increase in plasma NEFA upregulates the Toll-like receptor network in human muscle. Diabetologia. 2014 Mar;57(3):582-91. doi: 10.1007/s00125-013-3111-x. Epub 2013 Dec 14. PMID 24337154

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 of 52 participants were randomized. Of those not randomized, 40 did not meet inclusion criteria.
Groups:
- Lipid Then Saline: Intralipid 20% 30 ml/h for 48 h, then saline 30 ml/h for 48 h
- Saline Then Lipid: Saline infusion 30 ml/h for 48 h, then lipid 30 ml/h for 48 h
Period: First Intervention (48 h)
Arm/Group | Lipid Then Saline | Saline Then Lipid
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0
Period: Washout (4-6 Weeks)
Arm/Group | Lipid Then Saline | Saline Then Lipid
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0
Period: Second Intervention (48 h)
Arm/Group | Lipid Then Saline | Saline Then Lipid
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either lipid or saline
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Muscle Insulin Sensitivity-M Value
Description: Forty eight hrs after lipid or saline infusion, muscle insulin sensitivity will be measured by insulin clamp. The results are compared to determine whether lipid infusion reduces muscle insulin sensitivity compared to saline infusion..
  The M value is defined as the exogenous glucose infusion rate at steady state (i.e, when the exogenous glucose infusion rate is equal to the rate of whole body glucose disposal).
Time Frame: 48 hr after lipid/saline infusion
Measure: Mean (Standard Error); unit: mg/kg.min
Groups:
- Saline: Saline infusion at 30 ml/h for 48 h
- Intralipid: liposyn infusion at 30 ml/h for 48 hrs
Arm/Group | Saline | Intralipid
Number analyzed (Participants) | 12 | 12
mg/kg.min | 9.9 (0.7) | 8.3 (0.7)

2. Secondary Outcome: TLR4 Messenger Ribonucleic Acid (mRNA) in Muscle
Description: Forty eight hrs after lipid or saline infusion, muscle TLR4 mRNA levels will be measured by RT-PCR. The results are compared to determine whether lipid infusion increases muscle TLR4 mRNA expression compared to saline infusion.
  Saline mean was used to normalize the data for both arms.
Time Frame: 48 hr following lipid/saline infusion, pre-clamp
Measure: Mean (Standard Error); unit: ng TLR4 mRNA/ng Actin mRNA
Arm/Group | Saline | Intralipid
Number analyzed (Participants) | 12 | 12
ng TLR4 mRNA/ng Actin mRNA | 1 (0.15) | 1.6 (0.2)

3. Secondary Outcome: Extracellular Signal-regulated Kinase (ERK) Phosphorylation in Muscle
Description: Forty eight hrs after lipid or saline infusion, muscle ERK phosphorylation will be measured by western blot. The results are compared to determine whether lipid infusion increases muscle ERK phosphorylation compared to saline infusion. Saline mean was used to normalize the data for both arms.
Time Frame: 48 hr following lipid or saline infusion, pre-clamp
Measure: Mean (Standard Error); unit: densitometry value
Arm/Group | Saline | Intralipid
Number analyzed (Participants) | 12 | 12
densitometry value | 1.0 (0.18) | 1.95 (0.3)

ADVERSE EVENTS:
Groups:
- Saline: Intralipid infusion 20%, at 30 ml/h for 48 h, then washout 4-6 weeks, then saline 30 ml/h for 48 h
- Intralipid: Saline infusion 20%, at 30 ml/h for 48 h, then washout 4-6 weeks, then Intralipid 30 ml/h for 48 h
Arm/Group | Saline | Intralipid
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No